CLINICAL TRIAL: NCT02387502
Title: Comparative Evaluation of Macintosh, MacCoy and Airtraq Laryngoscope in Simulated Difficult Laryngoscopy Using Rigid Neck Collar
Brief Title: Comparison of Three Laryngoscopes in Difficult Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Bikramjit Das, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123-IEC/01/13
Record Dates: First submitted 2015-03-02; First posted 2015-03-13 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intubation with Macintosh laryngoscope (Experimental): 40 patients were intubated with Macintosh laryngoscope after simulating difficult laryngoscopy using rigid neck collar.
  Interventions: Device: Intubation- Macintosh laryngoscope
- Intubation with MacCoy laryngoscope (Active Comparator): 40 patients were intubated with MacCoy laryngoscope after simulating difficult laryngoscopy using rigid neck collar.
  Interventions: Device: Intubation- MacCoy laryngoscope
- Intubation with Airtraq laryngoscope (Active Comparator): 40 patients were intubated with Airtraq laryngoscope after simulating difficult laryngoscopy using rigid neck collar.
  Interventions: Device: Intubation- Airtraq laryngoscope

INTERVENTIONS:
Device: Intubation- Macintosh laryngoscope — Difficult intubation was simulated by using rigid neck collar. Then patients were intubated according to the assigned laryngoscopes. In Macintosh group, tip of the laryngoscope blade was placed in the vallecula and epiglottis was lifted. After visualization of the vocal cord, patients were intubated.
  Arms: Intubation with Macintosh laryngoscope
Device: Intubation- MacCoy laryngoscope — In MacCoy group, tip of the laryngoscope blade was placed in the vallecula and lever was pressed to flex the tip. After visualization of the vocal cord, patients were intubated.
  Arms: Intubation with MacCoy laryngoscope
Device: Intubation- Airtraq laryngoscope — In Airtraq group, the laryngoscope was loaded with endotracheal tube. Airtraq laryngoscope was inserted through midline and after visualization of image of vocal cord through its eyepiece, endotracheal tube was passed.
  Arms: Intubation with Airtraq laryngoscope

SUMMARY:
Tracheal intubation requires alignment of oro-pharyngeal-laryngeal axes. When these three axes are not aligned, intubation becomes difficult. In the researchers' study, the investigators simulated difficult laryngoscopy situation by using a rigid neck collar. This neck collar renders intubation difficult not only by restricting neck movement, but also reducing mouth opening. The investigators compared the performance of Macintosh, MacCoy and Airtraq laryngoscope in simulated difficult laryngoscopy using a rigid neck collar.

DETAILED DESCRIPTION:
Airtraq laryngoscope is an optical laryngoscope which allows visualization of vocal cord as a reflected image through multiple lenses and prisms. MacCoy laryngoscope is a modification of Macintosh laryngoscope. It has a lever which, when pressed, moves its flexible tip. In the investigators' study, the researchers compared the performances of Airtraq laryngoscope with MacCoy and Macintosh laryngoscopes in simulated difficult laryngoscopy using a rigid neck collar. The researchers recruited 120 patients and randomly divided those patients into three equal groups i.e. 30 patients in each group. These three groups are 1-Airtraq, 2-MacCoy and 3-Macintosh. The researchers compared efficacy and safety in these three laryngoscopes. The researchers compared efficacy in terms of time of intubation, ease of intubation, overall success, Intubation difficulty score, visualization of vocal cord in terms of POGO (percentage of Glottic Opening) score. The researchers compared safety in terms of hemodynamic pressor response and airway trauma.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II.
* Posted for elective surgery requiring general anesthesia and tracheal intubation

Exclusion Criteria:

* patients with anticipated difficult airway
* obese (body mass index (BMI)>30) patients
* patients with risk of pulmonary aspiration of gastric contents
* pregnant patients
* patients with airway distortion or trauma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Bhandari, M.D., Principal Investigator — Professor, Department of Anesthesiology, G.M.C. Haldwani

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 patients were recruited for the study. Recruitment process started in January 2014 and the study ended in December 2014. patients were recruited in the operating rooms of a tertiary care teaching hospital.
Pre-assignment Details: 30 patients were excluded from the study for not meeting the inclusion criteria.
Groups:
- Intubation With Macintosh Laryngoscope: After randomization, 40 patients were included in this group. After application of rigid neck collar, all patients were intubated with Macintosh laryngoscope. We observed and documented ease of intubation, time of intubation, overall success, number of attempts, Intubation Difficulty Score and POGO score. We also observed hemodynamic response in terms blood pressure and pulse rate. We assessed airway trauma after extubation.
  Intubation- Macintosh laryngoscope: Difficult intubation was simulated by using rigid neck collar. Then patients were intubated according to the assigned laryngoscopes. In Macintosh group, tip of the laryngoscope blade was placed in the vallecula and epiglottis was lifted. After visualization of the vocal cord, patients were intubated.
- Intubation With MacCoy Laryngoscope: After randomization, 40 patients were included in this group. After application of rigid neck collar, all patients were intubated with MacCoy laryngoscope. We observed and documented ease of intubation, time of intubation, overall success, number of attempts, Intubation Difficulty Score and POGO score. We also observed hemodynamic response in terms blood pressure and pulse rate. We assessed airway trauma after extubation.
  Intubation- MacCoy laryngoscope: In MacCoy group, tip of the laryngoscope blade was placed in the vallecula and lever was pressed to flex the tip. After visualization of the vocal cord, patients were intubated.
- Intubation With Airtraq Laryngoscope: After randomization, 40 patients were included in this group. After application of rigid neck collar, all patients were intubated with Airtraq laryngoscope. We observed and documented ease of intubation, time of intubation, overall success, number of attempts, Intubation Difficulty Score and POGO score. We also observed hemodynamic response in terms blood pressure and pulse rate. We assessed airway trauma after extubation.
  Intubation- Airtraq laryngoscope: In Airtraq group, the laryngoscope was loaded with endotracheal tube. Airtraq laryngoscope was inserted through midline and after visualization of image of vocal cord through its eyepiece, endotracheal tube was passed.
Period: Overall Study
Arm/Group | Intubation With Macintosh Laryngoscope | Intubation With MacCoy Laryngoscope | Intubation With Airtraq Laryngoscope
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubation With Macintosh Laryngoscope | Intubation With MacCoy Laryngoscope | Intubation With Airtraq Laryngoscope | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 40 | 120
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.35 (9.92) | 38.82 (9.62) | 35.47 (10.10) | 37.88 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 15 | 45
  Male | 26 | 24 | 25 | 75
Weight [Mean (Standard Deviation); unit: Kg] | 58.65 (6.03) | 58.62 (6.46) | 57.62 (5.65) | 58.30 (6.05)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.41 (1.11) | 22.43 (1.07) | 22.03 (1.13) | 22.29 (1.10)
Mallampati grade [Median (Inter-Quartile Range); unit: units on a scale] — The Mallampati classification is based on the structures visualized with maximal mouth opening and tongue protrusion in the sitting position.
  Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible.
  units on a scale | 2 [1 to 2] | 2 [1 to 2] | 1 [1 to 2] | 2 [1 to 2]
Thyromental distance [Mean (Standard Deviation); unit: cm] | 6.19 (0.40) | 6.16 (0.40) | 6.28 (0.44) | 6.21 (0.41)

OUTCOME MEASURES:

1. Primary Outcome: Time of Intubation
Description: Time of intubation is defined as the time from passing the device beyond the incisors to the confirmation of endotracheal tube placement by square wave capnograph tracings.
Time Frame: up to 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intubation With Macintosh Laryngoscope | Intubation With MacCoy Laryngoscope | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 40 | 40 | 40
seconds | 41.22 (4.72) | 37.62 (3.45) | 27.80 (3.87)

ADVERSE EVENTS:
Time Frame: up to 30 minutes after extubation
Arm/Group | Intubation With Macintosh Laryngoscope | Intubation With MacCoy Laryngoscope | Intubation With Airtraq Laryngoscope
Serious Adverse Events (participants affected / at risk) | 3/40 | 5/40 | 8/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intubation With Macintosh Laryngoscope (N=40) | Intubation With MacCoy Laryngoscope (N=40) | Intubation With Airtraq Laryngoscope (N=40)
Airway trauma (Injury, poisoning and procedural complications) | 3 | 5 | 8

LIMITATIONS AND CAVEATS:
The intubating anesthetist was not blind to the randomization of the laryngoscope. This could have led to bias. However, the primary outcome i.e. time of intubation was well defined and objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes